CLINICAL TRIAL: NCT04501809
Title: Vaginal Misoprostol Versus Combined Intracervical Foley's Catheter and Oxytocin Infusion for Second Trimester Pregnancy Termination in Women With Previous Caesarean Sections
Brief Title: Second Trimester Pregnancy Termination in Women With Previous Caesarean Sections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, basem mohamed hamed khalil, lecturer of obstetrics and gynecology/ MD ob/gyn / consultant of obstetrics and gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6276/14-7-2020
Record Dates: First submitted 2020-07-15; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Second Trimester Abortion
Keywords: abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Misoprostol group): (Active Comparator): seventy-nine patients will receive a loading dose of moistened misoprostol tablets ( Cytotec pfizer 400 mg) inserted vaginally and it will be followed by maintenance dose (200 mg) after six hours and repeated every 4 hours till the start of effective uterine contraction with maximum five doses in 24 hours duration .
  Interventions: Procedure: compare misoprostol with combined oxytocin and cervical foly catheter
- Group II (Combined group): (Active Comparator): seventy- nine patients will get intracervical Foleys Catheter insertion .a 16F (french units) Foley catheter will be introduced into the cervical canal to induce cervical ripping. The catheter will be fixed through inflation of the balloon with 30 milliliters of sterile solution when the catheter will be beyond the internal cervical os. After six hours of Foleys catheter fixation, we will start infusion of 10 international units (IU) of oxytocin on 500 ml ringer lactate by rate 125 ml\hr followed by one hour rest to allow diuresis. Increased gradually of oxytocin dose by 5 IU each time until achieving regular uterine contraction, maximum five doses in twenty -four hours duration.
  Interventions: Procedure: compare misoprostol with combined oxytocin and cervical foly catheter

INTERVENTIONS:
Procedure: compare misoprostol with combined oxytocin and cervical foly catheter — we will compare using misoprostol alone in one group with oxytocin and cervical catheter in the other group

SUMMARY:
it is a randomized controlled trial comparing the safety and efficacy of Vaginal Misoprostol versus combined Intracervical Foley's Catheter and Oxytocin Infusion for Second Trimester Pregnancy Termination. the patients will be sorted into 2 groups, Group I (Misoprostol group): seventy-nine patients and Group II (Combined group): seventy- nine patients. safety and efficacy of the procedure will be followed up and documented.

DETAILED DESCRIPTION:
Design: prospective randomized controlled trial Sitting: department of Obstetrics and Gynecology Faculty of Medicine, Zagazig University, Zagazig, Egypt Sample size calculation: thoroughly reviewing the use of vaginal misoprostol and intracervical Foleys catheter alone or in combination for mid trimester pregnancy termination, Rezk et al 2014 showed that the percentage of complications "fever and diarrhea" in the first group (misoprostol) was 30 % versus complications in the second group (intra cervical Foleys group)" cervical laceration "was 13.3 %. Therefore, at confidence level 95% and power 80%, using Epi info 7 the Sample size will be one hundred fifty-eight (158) patients.

Study participants: the study will include women indicated for termination of pregnancy between 14weeks-23 weeks and 6 days of gestation. The investigators will involve patients with a singleton pregnancy with one or multiple cesarean delivery. The investigators will exclude all patients with critical co-morbidities: bleeding disorders, chorioamnionitis, low-lying placenta, rupture uterus, myomectomy and contraindication to misoprostol or latex allergy. All women will undergo history taking, general examination, and local assessment for the cervix. Departmental US to confirm the diagnosis and indication for termination and position of the placenta. Blood tests will be done including blood group, full blood count matching, Antibodies screening and viral markers.

Randomization: After meeting eligibility criteria all participants will be counseled to the clinical trial. A signed documented consent form will be attached to their medical records. The patients will be sorted into two groups using a computerized random number generator in a sequence of sealed, numbered opaque envelopes, with a 1:1randomization ratio.

Group I (Misoprostol group): seventy-nine patients will receive a loading dose of moistened misoprostol tablets (cytotec pfizer 400 mg) inserted vaginally and it will be followed by maintenance dose (200 mg) after six hours and repeated every 4 hours till the start of effective uterine contraction with maximum five doses in 24 hours duration .

Group II (Combined group): seventy- nine patients will get intracervical Foleys Catheter insertion .Exposure of the cervix by means of a sterile speculum, a 16F Foley catheter will be introduced into the cervical canal to induce cervical ripping. The catheter will be fixed through inflation of the balloon with 30 milliliters of sterile solution when the catheter will be beyond the internal cervical os. Slight traction of the catheter will be exerted through tapping it to the inner thigh. After six hours of Foleys catheter fixation, The investigators will start infusion of 10 IU of oxytocin on 500 ml ringer lactate by rate 125 ml\hr followed by one hour rest to allow diuresis. Increased gradually of oxytocin dose by 5IU each time until achieving regular uterine contraction, maximum five doses in twenty -four hours duration. Therefore the maximum dose of oxytocin 100 IU over 24 hrs duration to avoid water intoxication.

Failed induction of abortion is considered if no fetal expulsion occurred within twenty for hours from the use of primary method of termination. The Demographic data and serial clinical monitoring will be recorded by the assigned on duty registrar.

ELIGIBILITY:
Inclusion Criteria:

* women indicated for termination of pregnancy between 14weeks-23 weeks and 6 days of gestation
* singleton pregnancy
* one or multiple cesarean delivery.

Exclusion Criteria:

* bleeding disorders
* chorioamnionitis
* low-lying placenta
* history of rupture uterus
* history of myomectomy
* contraindication to misoprostol

latex allergy.

Ages: 17 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
time to cervical dilatation in hours | 24 hours
  time between starting the medications and the real cervical dilatation
induction abortion interval in hours | 48 hours
  time between induction of abortion and expulsion of the products of conception
need for surgical evacuation | 48 hours
  some cases may be presented with retained products of conception with the need for surgical evacuation of the uterus

SECONDARY OUTCOMES:
sever hemorrhage | 48 hours
  comparing the prevalence of severe hemorrhage by postoperative hemoglobin percent in both groups.
patients satisfaction | 72 hours
  by patient written questionnaire about patient discomfort.
post-abortive infection | 7 days
  Number of participants with post-abortive infection is predicted by post-abortive C reactive protein (CRP) level
rupture uterus | 48 hours
  comparing the incidence of rupture uterus (clinically by sever abdominal pain and loss of uterine contractions and presence of free fluid by ultrasound) in both groups

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Zagazig University, Zagazig, East
  - Tolba Ewida Street, Zagazig, Sharqia Province

REFERENCES:
- [Derived] Elasy AN, Ibrahem MA, Elhawy LL, Hamed BM. Vaginal misoprostol versus combined intracervical foley's catheter and oxytocin infusion for second trimester pregnancy termination in women with previous caesarean sections: a randomised control trial. J Obstet Gynaecol. 2022 Oct;42(7):2962-2969. doi: 10.1080/01443615.2022.2118572. Epub 2022 Sep 23. PMID 36149628